CLINICAL TRIAL: NCT03958045
Title: Phase II Study of Combination Rucaparib With Nivolumab in Platinum-Sensitive Small Cell Lung Carcinoma Patients as Maintenance After Induction Therapy With Platinum Doublet
Brief Title: Combination Rucaparib With Nivolumab in Small Cell Lung Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhonglin Hao (Other)
Collaborators: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Zhonglin Hao, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49346 MCC-18-LUN-107-CLO
Record Dates: First submitted 2019-05-13; First posted 2019-05-21 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Small Cell Lung Cancer
Keywords: rucaparib; nivolumab; platinum-sensitive; maintenance; SCLC; immune checkpoint; PARP
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — rucaparib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Stage IV SCLC (Experimental): Patients with extensive stage (IV) SCLC (small cell lung cancer)
  Interventions: Combination Product: Rucaparib and Nivolumab

INTERVENTIONS:
Combination Product: Rucaparib and Nivolumab — Rucaparib (600mg BID) and Nivolumab (480mg IV q4 wk)

SUMMARY:
The purpose of this study is to evaluate survival and response rate of the combination rucaparib and nivolumab as maintenance therapy in platinum-sensitive small cell lung carcinoma.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is one of the most aggressive malignancies with a 5-year survival rate of less than 7%. SCLC is characterized by rapid doubling time, high growth fraction and early development of widespread metastases. SCLC accounts for roughly 93% of all high-grade neuroendocrine carcinomas. The prognosis for SCLC is extremely poor with a median survival less than a year for extensive-stage disease. Therapeutic options have not advanced significantly in over two decades, with frontline treatment consisting of platinum doublet therapy for 3-6 cycles. While most patients show an initial favorable response to Carboplatin/cisplatin + etoposide, this response is usually short-lived. Most patients relapse with resistant disease between 3 to 6 months after completion of initial chemotherapy.

Based on preclinical data supporting the role of immune checkpoint and PARP (poly ADP ribose polymerase ) inhibitors in SCLC, combining nivolumab and rucaparib has the potential to prolong progression-free survival and overall survival. These two classes of drugs have non-overlapping toxicities. This novel combination has not been tried in a front-line maintenance setting for SCLC.

Eligible patients will have pathological (biopsy) or cytologically confirmed stage IV SCLC, and have achieved either partial or complete response post frontline chemotherapy with platinum doublet. Patients will be treated with combination rucaparib and nivolumab. The recommended starting dose of rucaparib as a continuously administered oral monotherapy is 600 mg BID. Nivolumab will be administered as an intravenous infusion once every 4 weeks at a fixed dose of 480 mg. In the absence of treatment delays due to adverse event(s), treatment may continue for 24 months.

Progression-free survival, overall survival, disease control rates, objective response rate, quality of life, and tumor mutation burden will be evaluated during this study (up to 2 years).

ELIGIBILITY:
Inclusion Criteria

* Patients with histologically or cytologically confirmed stage IV, extensive stage, small cell lung cancer who achieved either partial or complete remission per RECIST 1.1 post frontline chemotherapy with platinum doublet (Cisplatin or Carboplatin/etoposide).
* Enrollment is within 6 weeks of last (4th cycle) of chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate Bone Marrow Function
* Adequate Hepatic Function

Exclusion Criteria

* Prior therapy with any antibody/drug targeting T-cell co-regulatory proteins (immune checkpoints)
* Major surgery within 4 weeks of initiation of study medication.
* Current use of (some) immunosuppressants
* Active infection requiring systemic therapy
* HIV/AIDS
* Hepatitis B virus or hepatitis C virus infection at screening
* Autoimmune disease
* Persisting toxicity related to prior therapy
* Pregnancy
* Vaccination (except inactive) within 4 weeks of the first dose of nivolumab
* Hypersensitivity to the study drugs
* Cardiovascular disease
* Untreated central nervous system (CNS) metastases or leptomeningeal carcinomatosis
* (Some) active secondary malignancy
* Active pneumonitis or interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhonglin Hao, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patients With Stage IV SCLC
Started | 33
Completed | 32
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Stage IV SCLC
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Duration (time) of progression-free survival after response to initial platinum-based therapy.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions from starting maintenance treatment
Time Frame: 0-2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Patients With Stage IV SCLC
Number analyzed (Participants) | 32
months | 11 [10 to 13]

2. Secondary Outcome: Disease Control Rate
Description: Disease control rate (DCR) is the number of patients who had either complete response (CR, Disappearance of all target lesions), partial response (PR, >=30% decrease in the sum of the longest diameter of target lesions) or stable disease (SD, less than 30% decrease in the sum of the biggest dimension but no more than 20% increase ) per RECICST 1.0 divided by the total number of patients. DOR= (CR+PR+SD)/Total number on trial x 100%.
  The timepoints were combined. The best responses were used in calculating disease control rate
Time Frame: 8 weeks, 16 weeks and 24 weeks post-treatment
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Stage IV SCLC
Number analyzed (Participants) | 33
percentage of participants | 33.3

3. Secondary Outcome: Overall Survival
Description: Percentage of surviving participants at 1 and 2 years
Time Frame: 0-2 years
Measure: Number; unit: percentage of participants
Arm/Group | Patients With Stage IV SCLC
Number analyzed (Participants) | 33
percentage of participants
  1 year | 93.55
  2 years | 52.82

4. Secondary Outcome: Objective Response Rate
Description: Objective response rate (ORR) is the proportion of patients with complete response or partial response according to RECIST v1.1. Patients with complete response at baseline will be excluded from ORR analysis.
  The timepoints were combined. The best responses were used in calculating objective response rate
Time Frame: 8 weeks, 16 weeks and 24 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Stage IV SCLC
Number analyzed (Participants) | 33
Participants | 4

5. Secondary Outcome: Quality of Life Scale Baseline
Description: Quality of life is assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) questionnaire, which probes function and symptoms. Scores range from 0-100. High scores on functional scales represent a high/healthy level of functioning; high scores symptom scales represent a high level of symptomology.
Time Frame: Baseline
Population: 3 participants did not answer all questions
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients With Stage IV SCLC
Number analyzed (Participants) | 32
units on a scale
  Physical Functioning | 76.1 (17)
  Role Functioning | 69.3 (27.8)
  Emotional Functioning: number analyzed (Participants) | 29
  Emotional Functioning | 78.1 (19.6)
  Cognitive Functioning: number analyzed (Participants) | 29
  Cognitive Functioning | 81 (22.6)
  Social Functioning: number analyzed (Participants) | 29
  Social Functioning | 72.4 (26.1)
  Global health status: number analyzed (Participants) | 29
  Global health status | 65.2 (17.7)

6. Secondary Outcome: Quality of Life Scale 4 Months
Description: as for outcome 5
Time Frame: 4 months
Population: Only 10 participants completed the scale at the 4 month timepoint
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients With Stage IV SCLC
Number analyzed (Participants) | 10
units on a scale
  Physical Functioning | 70.5 (14.7)
  Role Functioning | 65 (30.9)
  Emotional Functioning | 75.6 (24.1)
  Cognitive Functioning | 78.3 (26.1)
  Social Functioning | 73.3 (25.1)
  Global health status | 65.8 (14.4)

7. Secondary Outcome: Quality of Life Scale at Disease Progression
Description: as for outcome 5
Time Frame: Disease Progression up to 2 years
Population: Only 2 subjects have completed the questionnaire at progression. Due to this small sample size, the standard deviation can be 0 if the responses happen to be the same for questions related to "physical functioning"
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients With Stage IV SCLC
Number analyzed (Participants) | 2
units on a scale
  Physical Functioning | 66.7 (0)
  Role Functioning | 41.7 (35.4)
  Emotional Functioning | 45.8 (41.2)
  Cognitive Functioning | 41.7 (35.4)
  Social Functioning | 50 (23.6)
  Global health status | 50 (23.6)

8. Other Pre Specified Outcome: Tumor Mutation Burden
Description: Correlate tumor mutation burden with treatment response.
Time Frame: 0-3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: PD-L1 CPS
Description: A combined positive score (CPS) for Programmed Death Ligand 1 (PD-L1) will be derived from immunohistochemical analysis of tumor tissue.
Time Frame: 0-3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Patients With Stage IV SCLC
All-Cause Mortality (participants affected / at risk) | 16/33
Serious Adverse Events (participants affected / at risk) | 12/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Stage IV SCLC (N=33)
Anemia (Blood and lymphatic system disorders) | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flu like symptoms (General disorders) | 1
Enterocolitis infectious (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Stage IV SCLC (N=33)
Anemia (Blood and lymphatic system disorders) | 8
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 3
Blurred Vision (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 8
Mucositis Oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 10
Fatigue (General disorders) | 17
Fever (General disorders) | 2
Generalized Edema (General disorders) | 2
Pain (General disorders) | 3
Shingles (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Lung Infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 15
Alkaline phosphatase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 15
Blood bilirubin increased (Investigations) | 5
Creatinine increased (Investigations) | 7
Lymphocyte count decreased (Investigations) | 15
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 14
Thyroid stimulating hormone increased (Investigations) | 4
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 13
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Other (Respiratory, thoracic and mediastinal disorders) | 2
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT03958045/Prot_SAP_000.pdf